CLINICAL TRIAL: NCT04132934
Title: Observational Study Program Assessing Effectiveness and Tolerability of Gliclazide MR 60mg in Patients With Type 2 Diabetes Fasting During RAMADAN
Brief Title: Observational Study of Effectiveness and Tolerability of Gliclazide MR 60mg in Diabetic Patients Fasting During RAMADAN
Acronym: DIA-RAMADAN
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05762-004
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to assess effectiveness and tolerability of gliclazide MR 60mg during RAMADAN in a real world setting in 9 countries from Asia Pacific and Middle East/North Africa

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Male or female type 2 diabetic patients aged >18 years
* Patients with controlled or suboptimal controlled type 2 diabetes
* Patients with experience in SMBG controlling using glucometer
* Patients who are willing to fast during Ramadan
* Patients already treated with Gliclazide MR 60mg

Exclusion Criteria:

* Insulin therapy requirement
* Severe liver or renal failure
* HbA1c ≥ 9%
* Contraindication to gliclazide according to SmPC
* Pregnancy or breast feeding
* Previous experience of severe or repeated hypoglycemia events without triggered factor within the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes observing fast during Ramadan
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with at least one Hypoglycemia event | up to 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Medicales, Suresnes, France

REFERENCES:
- [Result] Hassanein M, Al Sifri S, Shaikh S, Abbas Raza S, Akram J, Pranoto A, Rudijanto A, Shaltout I, Fariduddin M, Mohd Izani Wan Mohamed W, Al Awadi F, Alessa T; DIA-RAMADAN study investigators. A real-world study in patients with type 2 diabetes mellitus treated with gliclazide modified-release during fasting: DIA-RAMADAN. Diabetes Res Clin Pract. 2020 May;163:108154. doi: 10.1016/j.diabres.2020.108154. Epub 2020 Apr 21. PMID 32330510
- [Derived] Hassanein M, Al Sifri S, Shaikh S, Raza SA, Akram J, Rudijanto A, Shaltout I, Fariduddin M, Mohamed WMIBW, Al Awadi F, Durocher A, Cortese V, Alessa T. Descriptive Regional Subanalysis of a Real-World Study in Patients with Type 2 Diabetes Treated with Gliclazide MR During Fasting: DIA-RAMADAN. Diabetes Ther. 2021 Jun;12(6):1703-1719. doi: 10.1007/s13300-021-01067-1. Epub 2021 May 11. PMID 33974216
- See also: A real-world study in patients with type 2 diabetes mellitus treated with gliclazide modified-release during fasting: DIA-RAMADAN. — https://www.ncbi.nlm.nih.gov/pubmed/32330510